CLINICAL TRIAL: NCT00673075
Title: Efficacy and Tolerability of Nebivolol Compared With Carvedilol in Patients With Coronary Artery Disease and Stage I or II Hypertension
Brief Title: The Effect of Nebivolol in Hypertensive Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: John Whalen, MD, Executive Director, Clinical Development, Cardiovascular, Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-06
Record Dates: First submitted 2008-04-29; First posted 2008-05-07 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Hypertension; Coronary Artery Disease
Keywords: carvedilol; Coreg (TM); hypertension; blood pressure; coronary artery disease; Nebivolol; BYSTOLIC (TM)
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — Nebivolol; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Encapsulated Nebivolol
  Interventions: Drug: Nebivolol
- 2 (Active Comparator): Encapsulated Carvedilol
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Nebivolol — Encapsulated Nebivolol 5 mg, 10 mg, 20, mg, 40 mg total daily dosage, oral administration once daily
  Other Names: Bystolic
  Arms: 1
Drug: Carvedilol — Encapsulated Carvedilol 12.5 mg, 25 mg, 50 mg total daily dosage, oral administration twice daily
  Other Names: Coreg
  Arms: 2

SUMMARY:
This study is being done to see if the blood pressure lowering effect of an approved drug nebivolol is comparable to that of another approved drug carvedilol for the treatment of hypertension in patients who have coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ambulatory outpatients 18 to 85 of age at screening
* Coronary artery disease as defined by: status post myocardial infarction (heart attack) greater than 14 days post event with no upper time limit (and followed by stress testing with additional imaging (echocardiographic or nuclear) within the 12 months prior to enrollment) and/or angiographic evidence of one or more major coronary arteries narrowing of greater than 50% and/or a history of percutaneous or surgical coronary revascularization greater than 4 months after that procedure at the time of enrollment.
* Qualifying blood pressure criteria for study entry and for randomization
* Willing to adhere to exercise stress (treadmill) tests

Exclusion Criteria:

* Unstable angina within 7 days of screening
* Potential coronary surgical/intervention within the next 6 months
* Have any form of secondary hypertension
* Have a history of hypersensitivity to nebivolol, metoprolol, carvedilol, or any beta blocker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Lukic, MD., M.Sc, Study Director — Forest Research Institute, Inc., a Subsidiary of Forest Laboratories, Inc.
Locations (33):
- United States (33):
  - Forest Investigative Site, Birmingham, Alabama
  - Forest Investigative Site, Peoria, Arizona
  - Forest Investigative Site, Buena Park, California
  - Forest Investigative Site, Los Angeles, California
  - Forest Investigative Site, Orange, California
  - Forest Investigator Site, Santa Ana, California
  - Forest Investigative Site, Guilford, Connecticut
  - Forest Investigator Site, Coral Gables, Florida
  - Forest Investigative Site, Daytona Beach, Florida
  - Forest Investigator Site, Hollywood, Florida
  - Forest Investigator Site, New Smyrna Beach, Florida
  - Forest Investigative Site, Orlando, Florida
  - Forest Investigator Site, Winter Haven, Florida
  - Forest Investigative Site, Chicago, Illinois
  - Forest Investigator Site, Indianapolis, Indiana
  - Forest Investigator Site, Lafayette, Louisiana
  - Forest Investigator Site, Auburn, Maine
  - Forest Investigative Site, Pittsfield, Massachusetts
  - Forest Investigator Site, Worcester, Massachusetts
  - Forest Investigative Site, Detroit, Michigan
  - Forest Investigative Site, Lansing, Michigan
  - Forest Investigator Site, Las Vegas, Nevada
  - Forest Investigative Site, Northport, New York
  - Forest Investigative Site, The Bronx, New York
  - Forest Investigative Site, Charlotte, North Carolina
  - Forest Investigator Site, Lenoir, North Carolina
  - Forest Investigative Site, Fargo, North Dakota
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Lancaster, Pennsylvania
  - Forest Investigative Site, Charleston, South Carolina
  - Forest Investigator Site, Florence, South Carolina
  - Forest Investigative Site, Cleveland, Tennessee
  - Forest Investigative Site, Carrollton, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was April 2008 to May 2009 at 35 US locations.
Pre-assignment Details: All patients went through a 4-week, single blind, metoprolol run-in phase before randomization.
Groups:
- Nebivolol: Encapsulated Nebivolol
- Carvedilol: Encapsulated Carvedilol
Period: Overall Study
Arm/Group | Nebivolol | Carvedilol
Started | 21 | 18
Completed | 12 | 11
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Carvedilol | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 9 | 9 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.5) | 66.6 (10.3) | 63.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 20 | 12 | 32
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Diastolic Blood Pressure (DBP)
Description: Peripheral diastolic blood pressure (DBP) at post-baseline (visit 13, week 18)
Time Frame: 18 weeks post initiation of randomized treatment
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Nebivolol | Carvedilol
Number analyzed (Participants) | 13 | 12
mmHg
  Baseline | 81.1 (1.7) | 78.2 (1.8)
  Post-baseline | 78.0 (2.4) | 79.3 (2.6)

2. Secondary Outcome: Peripheral Systolic Blood Pressure (SBP)
Description: Peripheral systolic blood pressure (SBP) at visit 13 (week 18)
Time Frame: 18 weeks post initiation of randomized treatment
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Nebivolol | Carvedilol
Number analyzed (Participants) | 13 | 12
mmHg
  Baseline | 135.1 (2.5) | 136.9 (2.4)
  Post-Baseline | 129.6 (3.7) | 137.3 (4.4)

3. Secondary Outcome: Proportion of Patients With Peripheral SBP <140 mm Hg and DBP <90 mm Hg at Week 18
Description: Proportion of Patients with Peripheral SBP <140 mm Hg and DBP <90 mm Hg at Week 18
Time Frame: 18 weeks post-treatment
Measure: Number; unit: participants
Arm/Group | Nebivolol | Carvedilol
Number analyzed (Participants) | 13 | 12
participants | 11 | 5

4. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) (%) at Week 18
Description: Left ventricular ejection fraction (LVEF) (%) at Week 18
Time Frame: 18 weeks post-treatment
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Nebivolol | Carvedilol
Number analyzed (Participants) | 12 | 12
percentage
  Baseline | 61.43 (0.562) | 60.442 (1.125)
  Post baseline | 61.93 (0.503) | 60.775 (0.614)

ADVERSE EVENTS:
Time Frame: The adverse event reporting timeframe was 16 months - from June,2008 until October, 2009.
Groups:
- Nebivolol Combined Up-Titration and Stable-dose: Encapsulated Nebivolol Combined Up-Titration and Stable-Dose Periods
- Carvedilol Combined Up-Titration and Stable-dose: Encapsulated Carvedilol Combined Up-Titration and Stable-Dose Periods
- Nebivolol Down-Titration: Encapsulated Nebivolol Down-Titration Period
- Carvedilol Down-Titration: Encapsulated Carvedilol Down-Titration Period
Arm/Group | Nebivolol Combined Up-Titration and Stable-dose | Carvedilol Combined Up-Titration and Stable-dose | Nebivolol Down-Titration | Carvedilol Down-Titration
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/18 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 9/21 | 10/18 | 1/12 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol Combined Up-Titration and Stable-dose (N=21) | Carvedilol Combined Up-Titration and Stable-dose (N=18) | Nebivolol Down-Titration (N=12) | Carvedilol Down-Titration (N=11)
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol Combined Up-Titration and Stable-dose (N=21) | Carvedilol Combined Up-Titration and Stable-dose (N=18) | Nebivolol Down-Titration (N=12) | Carvedilol Down-Titration (N=11)
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Painful defaecatio (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Tinea infecton (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early because of difficulties with enrollment. Only 39 out of 160 planned patients were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 60 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential information. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in the publication. On sponsor's request, PI shall delay submission for any pub while sponsor files patent applications. Any publication will give recognition to Sponsor's support.